CLINICAL TRIAL: NCT04091321
Title: Association Between Chronic Headache and Back Pain With Childbirth
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Pamela Flood, Professor, Stanford University
Other Study IDs: 52732
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Headache Disorders, Secondary; Post-Dural Puncture Headache; Migraine Disorders; Back Pain; Anesthesia
MeSH Terms: conditions — Headache Disorders, Secondary; Post-Dural Puncture Headache; Migraine Disorders; Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Headache: Women who endorse chronic headache
- Chronic Back Pain: Women who endorse chronic back pain

SUMMARY:
This study uses a single questionnaire to evaluate two separate primary outcomes:

1. To identify association between chronic headache in women who have given birth to children as compared to a control group of women who have raised children but have not given birth to them
2. To identify association between chronic back pain in women who have given birth to children as compared to a control group of women who have raised children but have not given birth to them

DETAILED DESCRIPTION:
Chronic headache and back pain have an excess prevalence in women as compared to men. This study uses a single survey that uses logic to assess for association between childbirth and chronic headache and between childbirth and chronic back pain using screening questions. The questions are, "Do you suffer from chronic headaches" and "Do you suffer from chronic back pain". Depending on the answer to the screening question, the subject will be given further questions only related to the syndrome that they endorsed.

Arm 1) There is an association between chronic headache and childbirth over and above raising children. Secondary outcomes are temporal association between onset or worsening of headache and childbirth, association between migraine headache and childbirth, association between chronic headache and anesthetic complications.

Arm 2) There is an association between chronic back pain and childbirth over and above raising children. Secondary outcomes are temporal association between onset or worsening of back pain and childbirth, association between chronic headache and anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Female representation

Exclusion Criteria:

* None

Min Age: 10 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Study Population: Chronic pain patients who have elected to be contacted for research studies
Sampling Method: Non-Probability Sample
Enrollment: 1112 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Chronic headache | 10 minute questionnaire
  Percent of patients with chronic headache who gave birth to children/Percent of patients with chronic headache who raised children but did not gave birth
Chronic back pain | 10 minute questionnaire
  Percent of patients with chronic back pain who gave birth to children/Percent of patients with chronic back pain who did not gave birth

SECONDARY OUTCOMES:
Migraine | 10 minute questionnaire
  Percent of patients with migraine who gave birth to children/Percent of patients with migraine who did not gave birth
Temporal coincidence of headache and childbirth | 10 minute questionnaire
  Women who developed or had worse headache within one year of delivery compared to one year of starting to raise a child not delivered
Temporal coincidence of headache and dural puncture | 10 minute questionnaire
  Women who developed or had worse headache within one year of dural puncture compared to those who did not have a dural puncture

OTHER OUTCOMES:
Temporal coincidence of back pain and regional anesthesia | 10 minute questionnaire
  Women who developed or had worse back pain within one year of regional anesthesia compared to those who did not have regional anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Depending on agreement. De identified data only

REFERENCES:
- [Derived] Zhang M, Cooley C, Ziadni MS, Mackey I, Flood P. Association between history of childbirth and chronic, functionally significant back pain in later life. BMC Womens Health. 2023 Jan 3;23(1):4. doi: 10.1186/s12905-022-02023-2. PMID 36597120